CLINICAL TRIAL: NCT02742766
Title: A Phase I, Randomized, Placebo-Controlled, Double-Blind (Sponsor Unblind), Three Part Study to Evaluate the Safety, Tolerability, Preliminary PK and PD of Single and Repeat Oral Doses of GSK3008356 in Healthy Subjects and Obese Subjects
Brief Title: Safety, Tolerability and Preliminary Pharmacokinetics (PK) and Pharmacodynamics (PD) of Single and Repeat Oral Doses of GSK3008356 in Healthy and Obese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Collaborators: Nucleus Network Ltd (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 204856
Record Dates: First submitted 2016-03-10; First posted 2016-04-19 (Estimated); Results first posted 2019-01-15 (Actual); Last update posted 2019-07-24 (Actual); Status verified 2019-07

CONDITIONS: Healthy Volunteers
Keywords: Dose escalation study; Safety; Pharmacodynamics; Pharmacokinetics; GSK3008356; Tolerability
MeSH Terms: interventions — GSK3008356

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Part 1 - GSK3008356 single dose and multiple doses (Experimental): Healthy subjects will receive GSK3008356 in morning as single dose or multiple doses of 5 milligrams (mg), 10 mg, 30 mg,45 mg, 75 mg, 90 mg, 125, 180 mg, 200 mg, 250 mg total daily dose or matching placebo in eleven sequential cohorts while receiving a standard fat meal. The initial dosing for the first cohort will be staggered so that 2 subjects will be dosed as sentinel subjects. Provided there are no safety concerns, the remainder of the subjects scheduled for the cohort may be dosed. Eight subjects will be enrolled in each cohort.
  Interventions: Drug: GSK3008356; Drug: Placebo
- Part 2 - GSK3008356 14 day repeat dose (Experimental): Healthy subjects will receive GSK3008356 or matching placebo, as 14 daily doses in the three sequential cohorts. Subjects in cohort 1 will receive their daily dose in morning, while subjects in cohort 2 and cohort 3 will receive their daily dose in evening. In all the three cohorts, Day 1 and day 14 dosing will occur while receiving a standard fat meal in morning. Eight subjects will be enrolled in each cohort.
  Interventions: Drug: GSK3008356; Drug: Placebo
- Part 3 - GSK3008356 28 day repeat dose (Experimental): Obese subjects will receive GSK3008356 or matching placebo, as 28 daily doses in the three parallel cohorts. Cohort 1 will evaluate 1 dose strength of GSK3008356 (or matching placebo) administered as morning doses. Cohorts 2 and 3 will evaluate 2 dose strengths (1 per cohort) of GSK3008356 (or matching placebo) administered in the evening. Ten subjects will be enrolled in each cohort.
  Interventions: Drug: GSK3008356; Drug: Placebo

INTERVENTIONS:
Drug: GSK3008356 — This intervention is available as 0.5, 1, 5, and 25 mg white oral tablet. The formulation will be used to administer dose of 5 mg, 10 mg, 30 mg, 45 mg, 75 mg, 90 mg, 125 mg, 180 mg, 200 mg, and 250 mg total daily dose during the study.
Drug: Placebo — This intervention is available as white oral tablet. The formulation will be used as a matching placebo for GSK3008356 during the study.

SUMMARY:
This study is a phase I, randomized, placebo-controlled, double-blind (sponsor unblind), three part study. The primary objective of the study is to characterize the safety, and tolerability of GSK3008356 single dose, 14 daily repeat doses in healthy subjects and 28 daily repeat doses in obese subjects. The study has three parts. Part 1, will be a single and multiple-dose, dose-rising study in healthy subjects. Part 2, will be a 14-day, repeat-dose, dose-rising study in healthy subjects, and part 3 will be a 28-day, repeat-dose study in obese subjects. For Parts 1 and 2, data from prior doses cohorts will be available prior to escalation decisions. Data from Parts 1 and 2 will be available prior to initiation of the three parallel cohorts in Part 3. A dose escalation meeting will be held to review these data and document the decision to proceed as planned or make any alterations in dosing, if indicated. Part 1, Part 2 and Part 3 study will have approximately 88, 24 and 30 subjects, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 65 years of age inclusive, at the time of signing the informed consent.
* For Part 1 and Part 2: Healthy as determined by the investigator or medically qualified designee based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring.
* For Part 3: Obese subjects may have chronic disease not specifically excluded and not requiring chronic medication for treatment and are otherwise healthy as determined by the investigator or medically qualified designee based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring. A subject with a clinical abnormality or laboratory parameter(s) which is/are not specifically listed in the inclusion or exclusion criteria, outside the reference range for the population being studied may be included only if the investigator in consultation with the Medical Monitor agree and document that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Body weight >=50 kilograms (kg)
* For Part 1 and Part 2 body mass index (BMI) 19-25 kilogram per meter square (inclusive)
* For Part 3 BMI >=30 kilogram per meter square
* Males or Females of non-childbearing potential as follows: Male subjects with female partners of child bearing potential must comply with the following contraception requirements from the time of first dose of study medication until at least five half-lives of study medication after the last dose of study medication.

  1. Vasectomy with documentation of azoospermia.
  2. Male condom plus partner use of one of the following contraceptive options: Contraceptive subdermal implant; Intrauterine device or intrauterine system; Oral Contraceptive, either combined or progestogen alone; Injectable progestogen; Contraceptive vaginal ring; Percutaneous contraceptive patches
* Males or Females of non-childbearing potential as follows: A female subject is eligible to participate if she is not pregnant (as confirmed by a negative serum human chorionic gonadotrophin [hCG] test), not lactating, and the following condition applies:

Non-reproductive potential defined as: Pre-menopausal females with one of the following: Documented tubal ligation; Documented hysteroscopic tubal occlusion procedure with follow-up confirmation of bilateral tubal occlusion; Hysterectomy; Documented Bilateral Oophorectomy. Postmenopausal defined as 12 months of spontaneous amenorrhea in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) > 40 milli-international units per milliliter (MlU/ml) and estradiol < 40 picograms (pg) per ml (<147 picomoles per liter (pmol/L) is confirmatory. Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will not be allowed.

The investigator is responsible for ensuring that subjects understand how to properly use these methods of contraception.

* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the consent form and in this protocol.

Exclusion Criteria:

* Alanine aminotransferase (ALT) and bilirubin >1.5 times upper limit of normal (isolated bilirubin >1.5 times upper limit of normal is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones)
* QTcF >450 millisecond (msec)
* Current or chronic history of gastrointestinal illness or conditions interfering with normal gastrointestinal anatomy or motility. Examples include gastrointestinal bypass surgery, cholecystectomy, partial or total gastrectomy, small bowel resection, vagotomy, malabsorption, Crohn's disease, ulcerative colitis, irritable bowel syndrome (IBS), or celiac sprue.
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study drug, unless in the opinion of the Investigator and GlaxoSmithKline (GSK) Medical Monitor the medication will not interfere with the study procedures or compromise subject safety. By exception, subject may take acetaminophen (<=2 grams per day) up to 48 hours prior to the first dose of study drug.
* Subjects should refrain from consumption of red wine, Seville oranges, grapefruit or grapefruit juice and/or pummelos, exotic citrus fruits, grapefruit hybrids or fruit juices from 7 days prior to the first dose of study medication until after the final dose.
* History of regular alcohol consumption within 6 months of the study defined as an average weekly intake of >14 standard drinks. One standard drink is equivalent to 10 grams of alcohol: 285 milliliter (mL) of beer, 100 mL of wine or 30 mL of 40% alcohol by volume distilled spirits.
* For Part 1 and Part 2, urinary cotinine levels indicative of smoking or history or regular use of tobacco- or nicotine-containing products within 3 months prior to screening.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or Medical Monitor, contraindicates their participation.
* Presence of hepatitis B surface antigen (HBsAg), positive hepatitis C antibody test result at screening or within 3 months prior to first dose of study treatment. For potent immunosuppressive agents, subjects with presence of hepatitis B core antibody (HBcAb) should also be excluded.
* A positive pre-study drug/alcohol screen.
* A positive test for human immunodeficiency virus (HIV) antibody.
* Where participation in the study would result in donation of blood or blood products in excess of 750 mL within 90 day period.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2016-03-14 (Actual); Primary Completion 2017-06-16 (Actual); Study Completion 2017-06-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://www.clinicalstudydatarequest.com/SearchAllPostings.aspx?searchparam=204856

REFERENCES:
- [Background] Okour M, Gress A, Zhu X, Rieman D, Lickliter JD, Brigandi RA. First-in-Human Pharmacokinetics and Safety Study of GSK3008356, a Selective DGAT1 Inhibitor, in Healthy Volunteers. Clin Pharmacol Drug Dev. 2019 Nov;8(8):1088-1099. doi: 10.1002/cpdd.691. Epub 2019 Apr 5. PMID 30950565

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 104 participants (80 in Part 1 and 24 in Part 2) were randomized to receive either study medication or placebo. This study was conducted at a single center in Australia from 14-March-2016 to 16-June-2017.
Pre-assignment Details: This study was planned to be conducted in 3 parts: Part 1 (single-day dosing) and Part 2 (repeat dose) dose-rising study in healthy participants and Part 3 (repeat dose) in obese participants. Part 3 was not conducted since a tolerable dose with sufficient pharmacodynamic effects was not identified in Part 2 due to gastrointestinal issues.
Groups:
- Part 1- Placebo: Eligible participants received GSK3008356 matching placebo tablets via oral route (as either single or multiple doses) along with a 30% fat by calorie meal approximately 2 hours after the morning dose for a single day.
- Part 1-Cohort A1: GSK3008356 5 mg: Eligible participants received a single morning dose of GSK3008356 tablets via oral route (total dose of 5 milligrams [mg]) along with a 30% fat by calorie meal approximately 2 hours after the morning dose.
- Part 1-Cohort A2: GSK3008356 10 mg: Eligible participants received a single morning dose of GSK3008356 tablets via oral route (total dose of 10 mg) along with a 30% fat by calorie meal approximately 2 hours after the morning dose.
- Part 1-Cohort A3: GSK3008356 30 mg: Eligible participants received a single morning dose of GSK3008356 tablets via oral route (total dose of 30 mg) along with a 30% fat by calorie meal approximately 2 hours after the morning dose.
- Part 1-Cohort A4: GSK3008356 75 mg: Eligible participants received a single morning dose of GSK3008356 tablets via oral route (total dose of 75 mg) along with a 30% fat by calorie meal approximately 2 hours after the morning dose.
- Part 1-Cohort A5: GSK3008356 200 mg: Eligible participants received a single morning dose of GSK3008356 tablets via oral route (total dose of 200 mg) along with a 30% fat by calorie meal approximately 2 hours after the morning dose.
- Part 1-Cohort A6: GSK3008356 125 mg: Eligible participants received a single morning dose of GSK3008356 tablets via oral route (total dose of 125 mg) along with a 30% fat by calorie meal approximately 2 hours after the morning dose.
- Part 1-Cohort A7: GSK3008356 100 mg (0 h, 4 h): Eligible participants received GSK3008356 tablets via oral route (total dose of 200 mg such that one 100 mg dose was administered at 0 hour [h] and 4 h) along with a 30% fat by calorie meal approximately 2 hours after the morning dose in a single day.
- Part 1-Cohort A8: GSK3008356 100 mg (0 h, 16 h): Eligible participants received GSK3008356 tablets via oral route (total dose of 200 mg such that one 100 mg dose was administered at 0 h and 16 h) along with a 30% fat by calorie meal approximately 2 hours after the morning dose in a single day.
- Part 1-Cohort A9: GSK3008356 200 mg Evening Dose: Participants in this arm were planned to receive a single evening dose of GSK3008356 tablets via oral route (total dose of 200 mg) along with a 30% fat by calorie meal approximately 2 hours after the evening dose; but this arm was cancelled.
- Part 1-Cohort A10: GSK3008356 10 mg q1h x 9 Doses: Eligible participants received GSK3008356 tablets via oral route (total dose of 90 mg such that a 10 mg dose was administered once every hour [q1h] for a total of 9 doses) along with a 30% fat by calorie meal approximately 2 hours after the first morning dose in a single day.
- Part 1-Cohort A11: GSK3008356 5 mg q1h x 9 Doses: Eligible participants received GSK3008356 tablets via oral route (total dose of 45 mg such that a 5 mg dose was administered q1h for a total of 9 doses) along with a 30% fat by calorie meal approximately 2 hours after the first morning dose in a single day.
- Part 2-Placebo: Eligible participants received GSK3008356 matching placebo tablets via oral route (repeat doses) for a period of 14 days. Day 1 and Day 14 dosing occurred while receiving a standard 30% fat by calorie meal approximately 2 hours after the morning dose.
- Part 2-Cohort B1: GSK3008356 10 mg BID (0 h, 16 h): Eligible participants received GSK3008356 tablets twice-daily (BID) via oral route (total daily dose of 20 mg such that a 10 mg dose was administered at 0 h and 16 h) for a period of 14 days. Day 1 and Day 14 dosing occurred while receiving a standard 30% fat by calorie meal approximately 2 hours after the morning dose.
- Part 2-Cohort B2: GSK3008356 1 mg BID (0 h, 16 h): Eligible participants received GSK3008356 tablets BID via oral route (total daily dose of 2 mg such that a 1 mg dose was administered at 0 h and 16 h) for a period of 14 days. Day 1 and Day 14 dosing occurred while receiving a standard 30% fat by calorie meal approximately 2 hours after the morning dose.
- Part 2-Cohort B3: GSK3008356 3 mg BID (0 h, 16 h): Eligible participants received GSK3008356 tablets BID via oral route (total daily dose of 6 mg such that a 3 mg dose was administered at 0 h and 16 h) for a period of 14 days. Day 1 and Day 14 dosing occurred while receiving a standard 30% fat by calorie meal approximately 2 hours after the morning dose.
- Part 3: Obese Participants Cohort 1: Participants in this arm were planned to receive 28 daily doses so as to evaluate 1 dose strength of GSK3008356 (or matching placebo) administered as morning doses. Part 3 was not conducted since a tolerable dose with sufficient pharmacodynamic effects was not identified in Part 2 due to gastrointestinal issues.
- Part 3: Obese Participants Cohort 2; Part 3: Obese Participants Cohort 3: Participants in this arm were planned to receive 28 daily doses so as to evaluate 1 dose strength of GSK3008356 (or matching placebo) administered as evening doses. Part 3 was not conducted since a tolerable dose with sufficient pharmacodynamic effects was not identified in Part 2 due to gastrointestinal issues.
Period: Part 1 (Up to 8 Days)
Arm/Group | Part 1- Placebo | Part 1-Cohort A1: GSK3008356 5 mg | Part 1-Cohort A2: GSK3008356 10 mg | Part 1-Cohort A3: GSK3008356 30 mg | Part 1-Cohort A4: GSK3008356 75 mg | Part 1-Cohort A5: GSK3008356 200 mg | Part 1-Cohort A6: GSK3008356 125 mg | Part 1-Cohort A7: GSK3008356 100 mg (0 h, 4 h) | Part 1-Cohort A8: GSK3008356 100 mg (0 h, 16 h) | Part 1-Cohort A9: GSK3008356 200 mg Evening Dose | Part 1-Cohort A10: GSK3008356 10 mg q1h x 9 Doses | Part 1-Cohort A11: GSK3008356 5 mg q1h x 9 Doses | Part 2-Placebo | Part 2-Cohort B1: GSK3008356 10 mg BID (0 h, 16 h) | Part 2-Cohort B2: GSK3008356 1 mg BID (0 h, 16 h) | Part 2-Cohort B3: GSK3008356 3 mg BID (0 h, 16 h) | Part 3: Obese Participants Cohort 1 | Part 3: Obese Participants Cohort 2 | Part 3: Obese Participants Cohort 3
Started | 20 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 0 | 6 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 20 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 0 | 6 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 2 (Up to 22 Days)
Arm/Group | Part 1- Placebo | Part 1-Cohort A1: GSK3008356 5 mg | Part 1-Cohort A2: GSK3008356 10 mg | Part 1-Cohort A3: GSK3008356 30 mg | Part 1-Cohort A4: GSK3008356 75 mg | Part 1-Cohort A5: GSK3008356 200 mg | Part 1-Cohort A6: GSK3008356 125 mg | Part 1-Cohort A7: GSK3008356 100 mg (0 h, 4 h) | Part 1-Cohort A8: GSK3008356 100 mg (0 h, 16 h) | Part 1-Cohort A9: GSK3008356 200 mg Evening Dose | Part 1-Cohort A10: GSK3008356 10 mg q1h x 9 Doses | Part 1-Cohort A11: GSK3008356 5 mg q1h x 9 Doses | Part 2-Placebo | Part 2-Cohort B1: GSK3008356 10 mg BID (0 h, 16 h) | Part 2-Cohort B2: GSK3008356 1 mg BID (0 h, 16 h) | Part 2-Cohort B3: GSK3008356 3 mg BID (0 h, 16 h) | Part 3: Obese Participants Cohort 1 | Part 3: Obese Participants Cohort 2 | Part 3: Obese Participants Cohort 3
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 6 | 6 | 6 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 6 | 5 (Day 4 study medication interrupted due to an AE and eventually withdrew from study on Day 5.) | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 6 | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 5 | 0 | 1 | 0 | 0 | 0
Period: Part 3 (Up to 36 Days)
Arm/Group | Part 1- Placebo | Part 1-Cohort A1: GSK3008356 5 mg | Part 1-Cohort A2: GSK3008356 10 mg | Part 1-Cohort A3: GSK3008356 30 mg | Part 1-Cohort A4: GSK3008356 75 mg | Part 1-Cohort A5: GSK3008356 200 mg | Part 1-Cohort A6: GSK3008356 125 mg | Part 1-Cohort A7: GSK3008356 100 mg (0 h, 4 h) | Part 1-Cohort A8: GSK3008356 100 mg (0 h, 16 h) | Part 1-Cohort A9: GSK3008356 200 mg Evening Dose | Part 1-Cohort A10: GSK3008356 10 mg q1h x 9 Doses | Part 1-Cohort A11: GSK3008356 5 mg q1h x 9 Doses | Part 2-Placebo | Part 2-Cohort B1: GSK3008356 10 mg BID (0 h, 16 h) | Part 2-Cohort B2: GSK3008356 1 mg BID (0 h, 16 h) | Part 2-Cohort B3: GSK3008356 3 mg BID (0 h, 16 h) | Part 3: Obese Participants Cohort 1 | Part 3: Obese Participants Cohort 2 | Part 3: Obese Participants Cohort 3
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Part 1, Cohort 9 was cancelled per emerging data that lowered the future no observed adverse event level (NOAEL) and made the dose level and strategy irrelevant. Part 3 was not conducted since a tolerable dose with sufficient pharmacodynamic effects was not identified in Part 2.
Groups:
- Part 1-Cohort A1: GSK3008356 5 mg: Eligible participants received a single morning dose of GSK3008356 tablets via oral route (total dose of 5 mg) along with a 30% fat by calorie meal approximately 2 hours after the morning dose.
- Part 1-Cohort A7: GSK3008356 100 mg BID (0 h, 4 h): Eligible participants received GSK3008356 tablets via oral route (total dose of 200 mg such that one 100 mg dose was administered at 0 h and 4 h) along with a 30% fat by calorie meal approximately 2 hours after the morning dose in a single day.
- Part 1-Cohort A8: GSK3008356 100 mg BID (0 h, 16 h): Eligible participants received GSK3008356 tablets via oral route (total dose of 200 mg such that one 100 mg dose was administered at 0 h and 16 h) along with a 30% fat by calorie meal approximately 2 hours after the morning dose in a single day.
- Part 1-Cohort A10: GSK3008356 10 mg q1h x 9 Doses: Eligible participants received GSK3008356 tablets via oral route (total dose of 90 mg such that a 10 mg dose was administered q1h for a total of 9 doses) along with a 30% fat by calorie meal approximately 2 hours after the first morning dose in a single day.
- Part 2-Cohort B1: GSK3008356 10 mg BID (0 h, 16 h): Eligible participants received GSK3008356 tablets BID via oral route (total daily dose of 20 mg such that a 10 mg dose was administered at 0 h and 16 h) for a period of 14 days. Day 1 and Day 14 dosing occurred while receiving a standard 30% fat by calorie meal approximately 2 hours after the morning dose.
- Total: Total of all reporting groups
Arm/Group | Part 1- Placebo | Part 1-Cohort A1: GSK3008356 5 mg | Part 1-Cohort A2: GSK3008356 10 mg | Part 1-Cohort A3: GSK3008356 30 mg | Part 1-Cohort A4: GSK3008356 75 mg | Part 1-Cohort A5: GSK3008356 200 mg | Part 1-Cohort A6: GSK3008356 125 mg | Part 1-Cohort A7: GSK3008356 100 mg BID (0 h, 4 h) | Part 1-Cohort A8: GSK3008356 100 mg BID (0 h, 16 h) | Part 1-Cohort A9: GSK3008356 200 mg Evening Dose | Part 1-Cohort A10: GSK3008356 10 mg q1h x 9 Doses | Part 1-Cohort A11: GSK3008356 5 mg q1h x 9 Doses | Part 2-Placebo | Part 2-Cohort B1: GSK3008356 10 mg BID (0 h, 16 h) | Part 2-Cohort B2: GSK3008356 1 mg BID (0 h, 16 h) | Part 2-Cohort B3: GSK3008356 3 mg BID (0 h, 16 h) | Part 3: Obese Participants Cohort 1 | Part 3: Obese Participants Cohort 2 | Part 3: Obese Participants Cohort 3 | Total
Number analyzed (Participants) | 20 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 0 | 6 | 6 | 6 | 6 | 6 | 6 | 0 | 0 | 0 | 104
Age, Continuous [Mean (Standard Deviation); unit: Years] | 24.8 (5.07) | 28.0 (16.49) | 25.8 (3.54) | 26.3 (4.46) | 26.0 (4.69) | 26.7 (5.65) | 24.3 (2.94) | 28.0 (7.04) | 31.5 (4.55) |  | 26.3 (4.76) | 24.7 (3.88) | 35.3 (12.75) | 26.5 (2.59) | 31.2 (11.51) | 25.8 (4.17) |  |  |  | 27.1 (7.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |  | 0 | 0 | 0 | 0 | 0 | 0 |  |  |  | 0
  Male | 20 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 |  | 6 | 6 | 6 | 6 | 6 | 6 |  |  |  | 104
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 3 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 2 |  | 2 | 1 | 0 | 0 | 0 | 1 |  |  |  | 12
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |  | 0 | 0 | 0 | 0 | 0 | 0 |  |  |  | 1
  White | 15 | 4 | 4 | 5 | 5 | 5 | 5 | 4 | 4 |  | 3 | 4 | 6 | 6 | 5 | 4 |  |  |  | 79
  Brazilian | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 |  | 0 | 0 | 0 | 0 | 0 | 0 |  |  |  | 2
  Chinese/Australian | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 |  | 0 | 0 | 0 | 0 | 0 | 0 |  |  |  | 1
  Egyptian/New Zealand | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |  | 0 | 0 | 0 | 0 | 0 | 0 |  |  |  | 1
  Half White Half Italian | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 |  | 0 | 0 | 0 | 0 | 0 | 0 |  |  |  | 1
  Indian | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |  | 0 | 0 | 0 | 0 | 0 | 0 |  |  |  | 1
  Latin | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |  | 1 | 1 | 0 | 0 | 0 | 0 |  |  |  | 2
  Moroccan | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 |  | 0 | 0 | 0 | 0 | 0 | 0 |  |  |  | 1
  Spanish/Jamaican/English/Irish | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 |  | 0 | 0 | 0 | 0 | 0 | 0 |  |  |  | 1
  Middle Eastern | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |  | 0 | 0 | 0 | 0 | 1 | 0 |  |  |  | 1
  South American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |  | 0 | 0 | 0 | 0 | 0 | 1 |  |  |  | 1

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Number of Participants With Abnormal Findings in Physical Examinations
Description: A complete physical examination included assessment of the cardiovascular, respiratory, gastrointestinal, dermatologic and neurological systems, height, and weight. Height was measured and recorded only at screening. A brief physical examination included assessments of the skin, lungs, cardiovascular system, and abdomen (liver and spleen). Weight was recorded with the brief physical exam, but was not part of the brief physical exam. Number of participants with abnormal findings in physical examinations in Part 1 are presented.
Time Frame: Up to Day 8
Population: Safety Population comprised of all participants who received at least one dose of study medication.
Measure: Number; unit: Participants
Groups:
- Part 1-Cohort A7: GSK3008356 100 mg (0 h, 4 h): Eligible participants received GSK3008356 tablets via oral route (total dose of 200 mg such that one 100 mg dose was administered at 0 h and 4 h) along with a 30% fat by calorie meal approximately 2 hours after the morning dose in a single day.
Arm/Group | Part 1- Placebo | Part 1-Cohort A1: GSK3008356 5 mg | Part 1-Cohort A2: GSK3008356 10 mg | Part 1-Cohort A3: GSK3008356 30 mg | Part 1-Cohort A4: GSK3008356 75 mg | Part 1-Cohort A5: GSK3008356 200 mg | Part 1-Cohort A6: GSK3008356 125 mg | Part 1-Cohort A7: GSK3008356 100 mg (0 h, 4 h) | Part 1-Cohort A8: GSK3008356 100 mg (0 h, 16 h) | Part 1-Cohort A9: GSK3008356 200 mg Evening Dose | Part 1-Cohort A10: GSK3008356 10 mg q1h x 9 Doses | Part 1-Cohort A11: GSK3008356 5 mg q1h x 9 Doses
Number analyzed (Participants) | 20 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 0 | 6 | 6
Participants | 2 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 |  | 0 | 0

2. Primary Outcome: Part 1: Number of Participants With Vital Signs of Potential Clinical Concern
Description: Vital signs included systolic and diastolic blood pressure and pulse rate and were measured with the participant in semi-supine position after 5 minutes rest. Temperature was also measured as a vital sign but did not require positioning or rest prior to measuring.
Time Frame: Up to Day 8
Population: Safety Population.
Measure: Number; unit: Participants
Arm/Group | Part 1- Placebo | Part 1-Cohort A1: GSK3008356 5 mg | Part 1-Cohort A2: GSK3008356 10 mg | Part 1-Cohort A3: GSK3008356 30 mg | Part 1-Cohort A4: GSK3008356 75 mg | Part 1-Cohort A5: GSK3008356 200 mg | Part 1-Cohort A6: GSK3008356 125 mg | Part 1-Cohort A7: GSK3008356 100 mg (0 h, 4 h) | Part 1-Cohort A8: GSK3008356 100 mg (0 h, 16 h) | Part 1-Cohort A9: GSK3008356 200 mg Evening Dose | Part 1-Cohort A10: GSK3008356 10 mg q1h x 9 Doses | Part 1-Cohort A11: GSK3008356 5 mg q1h x 9 Doses
Number analyzed (Participants) | 20 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 0 | 6 | 6
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 |  | 0 | 1

3. Primary Outcome: Part 1: Number of Participants With 12-lead Electrocardiogram (ECG) Values of Potential Clinical Concern
Description: Single 12-lead ECGs were obtained using an ECG machine that automatically calculated the heart rate and measured PR, QRS, and QT intervals, and QT interval corrected by Fridericia's formula (QTcF). Number of participants with 12-lead ECG values of potential clinical concern in Part 1 are presented.
Time Frame: Up to Day 4
Population: Safety Population.
Measure: Number; unit: Participants
Arm/Group | Part 1- Placebo | Part 1-Cohort A1: GSK3008356 5 mg | Part 1-Cohort A2: GSK3008356 10 mg | Part 1-Cohort A3: GSK3008356 30 mg | Part 1-Cohort A4: GSK3008356 75 mg | Part 1-Cohort A5: GSK3008356 200 mg | Part 1-Cohort A6: GSK3008356 125 mg | Part 1-Cohort A7: GSK3008356 100 mg (0 h, 4 h) | Part 1-Cohort A8: GSK3008356 100 mg (0 h, 16 h) | Part 1-Cohort A9: GSK3008356 200 mg Evening Dose | Part 1-Cohort A10: GSK3008356 10 mg q1h x 9 Doses | Part 1-Cohort A11: GSK3008356 5 mg q1h x 9 Doses
Number analyzed (Participants) | 20 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 0 | 6 | 6
Participants | 4 | 3 | 3 | 2 | 3 | 0 | 2 | 0 | 3 |  | 1 | 0

4. Primary Outcome: Part 1: Number of Participants With Clinically Significant Findings During Cardiac Monitoring
Description: Continuous lead II cardiac telemetry or cardiac monitoring was performed on Day 1. Number of participants with clinically significant findings during cardiac monitoring in Part 1 are presented.
Time Frame: Day 1
Population: Safety Population.
Measure: Number; unit: Participants
Arm/Group | Part 1- Placebo | Part 1-Cohort A1: GSK3008356 5 mg | Part 1-Cohort A2: GSK3008356 10 mg | Part 1-Cohort A3: GSK3008356 30 mg | Part 1-Cohort A4: GSK3008356 75 mg | Part 1-Cohort A5: GSK3008356 200 mg | Part 1-Cohort A6: GSK3008356 125 mg | Part 1-Cohort A7: GSK3008356 100 mg (0 h, 4 h) | Part 1-Cohort A8: GSK3008356 100 mg (0 h, 16 h) | Part 1-Cohort A9: GSK3008356 200 mg Evening Dose | Part 1-Cohort A10: GSK3008356 10 mg q1h x 9 Doses | Part 1-Cohort A11: GSK3008356 5 mg q1h x 9 Doses
Number analyzed (Participants) | 20 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 0 | 6 | 6
Participants | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 |  | 0 | 0

5. Primary Outcome: Part 1: Number of Participants With Laboratory Values of Potential Clinical Concern
Description: Hematology parameters included hematocrit, hemoglobin, platelets, white blood cells (WBC), neutrophils, lymphocytes, monocytes, eosinophils, basophils, mean corpuscular volume, mean corpuscular hemoglobin, mean corpuscular hemoglobin concentration, red blood cells (RBC) and reticulocytes. Clinical chemistry parameters included blood urea nitrogen, aspartate aminotransferase, alanine aminotransferase, gamma glutamyl transferase, alkaline phosphatase, uric acid, total protein, total and direct bilirubin, albumin, calcium, bile acids, chloride, creatinine, glucose (fasting/non-fasting), potassium, sodium and total carbon dioxide/bicarbonate. Urinalysis included specific gravity, potential of hydrogen (pH), glucose, protein, blood and ketones by dipstick and microscopic examination of urine (WBC, RBC and casts) within 120 minutes of collection.
Time Frame: Up to Day 8
Population: Safety Population.
Measure: Number; unit: Participants
Arm/Group | Part 1- Placebo | Part 1-Cohort A1: GSK3008356 5 mg | Part 1-Cohort A2: GSK3008356 10 mg | Part 1-Cohort A3: GSK3008356 30 mg | Part 1-Cohort A4: GSK3008356 75 mg | Part 1-Cohort A5: GSK3008356 200 mg | Part 1-Cohort A6: GSK3008356 125 mg | Part 1-Cohort A7: GSK3008356 100 mg (0 h, 4 h) | Part 1-Cohort A8: GSK3008356 100 mg (0 h, 16 h) | Part 1-Cohort A9: GSK3008356 200 mg Evening Dose | Part 1-Cohort A10: GSK3008356 10 mg q1h x 9 Doses | Part 1-Cohort A11: GSK3008356 5 mg q1h x 9 Doses
Number analyzed (Participants) | 20 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 0 | 6 | 6
Participants | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 |  | 0 | 1

6. Primary Outcome: Part 1: Number of Participants With Adverse Events (AE) and Serious Adverse Events (SAE)
Description: AE is any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product. For marketed medicinal products, this also includes failure to produce expected benefits (i.e., lack of efficacy), abuse or misuse. SAE is any untoward medical occurrence that, at any dose results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, or is a congenital anomaly/birth defect or is medically significant or is associated with liver injury and impaired liver function.
Time Frame: Up to Day 8
Population: Safety Population.
Measure: Number; unit: Participants
Arm/Group | Part 1- Placebo | Part 1-Cohort A1: GSK3008356 5 mg | Part 1-Cohort A2: GSK3008356 10 mg | Part 1-Cohort A3: GSK3008356 30 mg | Part 1-Cohort A4: GSK3008356 75 mg | Part 1-Cohort A5: GSK3008356 200 mg | Part 1-Cohort A6: GSK3008356 125 mg | Part 1-Cohort A7: GSK3008356 100 mg (0 h, 4 h) | Part 1-Cohort A8: GSK3008356 100 mg (0 h, 16 h) | Part 1-Cohort A9: GSK3008356 200 mg Evening Dose | Part 1-Cohort A10: GSK3008356 10 mg q1h x 9 Doses | Part 1-Cohort A11: GSK3008356 5 mg q1h x 9 Doses
Number analyzed (Participants) | 20 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 0 | 6 | 6
Participants
  AE | 5 | 2 | 1 | 1 | 3 | 4 | 4 | 3 | 3 |  | 0 | 4
  SAE | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |  | 0 | 0

7. Primary Outcome: Part 2: Number of Participants With Abnormal Findings in Physical Examination
Description: A complete physical examination included assessment of the cardiovascular, respiratory, gastrointestinal, dermatologic and neurological systems, height, and weight. Height was measured and recorded only at screening. A brief physical examination included assessments of the skin, lungs, cardiovascular system, and abdomen (liver and spleen). Weight was recorded with the brief physical exam, but was not part of the brief physical exam. Number of participants with abnormal findings in physical examinations in Part 2 are presented.
Time Frame: Up to Day 22
Population: Safety Population.
Measure: Number; unit: Participants
Arm/Group | Part 2-Placebo | Part 2-Cohort B1: GSK3008356 10 mg BID (0 h, 16 h) | Part 2-Cohort B2: GSK3008356 1 mg BID (0 h, 16 h) | Part 2-Cohort B3: GSK3008356 3 mg BID (0 h, 16 h)
Number analyzed (Participants) | 6 | 6 | 6 | 6
Participants | 2 | 2 | 3 | 4

8. Primary Outcome: Part 2: Number of Participants With Vital Signs of Potential Clinical Concern
Description: Vital signs included systolic and diastolic blood pressure and pulse and was measured with the participant in semi-supine position after 5 minutes rest. Temperature was also measured as a vital sign but did not require positioning or rest prior to measuring.
Time Frame: Up to Day 22
Population: Safety Population.
Measure: Number; unit: Participants
Arm/Group | Part 2-Placebo | Part 2-Cohort B1: GSK3008356 10 mg BID (0 h, 16 h) | Part 2-Cohort B2: GSK3008356 1 mg BID (0 h, 16 h) | Part 2-Cohort B3: GSK3008356 3 mg BID (0 h, 16 h)
Number analyzed (Participants) | 6 | 6 | 6 | 6
Participants | 1 | 0 | 0 | 1

9. Primary Outcome: Part 2: Number of Participants With 12-lead ECG Values of Potential Clinical Concern
Description: Single 12-lead ECGs were obtained using an ECG machine that automatically calculated the heart rate and measured PR, QRS, and QT intervals, and QTcF. Number of participants with 12-lead ECG values of potential clinical concern in Part 2 are presented.
Time Frame: Up to Day 17
Population: Safety Population.
Measure: Number; unit: Participants
Arm/Group | Part 2-Placebo | Part 2-Cohort B1: GSK3008356 10 mg BID (0 h, 16 h) | Part 2-Cohort B2: GSK3008356 1 mg BID (0 h, 16 h) | Part 2-Cohort B3: GSK3008356 3 mg BID (0 h, 16 h)
Number analyzed (Participants) | 6 | 6 | 6 | 6
Participants | 1 | 1 | 0 | 2

10. Primary Outcome: Part 2: Number of Participants With Clinically Significant Findings During Cardiac Monitoring
Description: Continuous lead II cardiac telemetry or cardiac monitoring was performed on Day 1. Number of participants with clinically significant findings during cardiac monitoring in Part 2 are presented.
Time Frame: Day 1 (Pre-dose to 4 hours post dose)
Population: Safety Population.
Measure: Number; unit: Participants
Arm/Group | Part 2-Placebo | Part 2-Cohort B1: GSK3008356 10 mg BID (0 h, 16 h) | Part 2-Cohort B2: GSK3008356 1 mg BID (0 h, 16 h) | Part 2-Cohort B3: GSK3008356 3 mg BID (0 h, 16 h)
Number analyzed (Participants) | 6 | 6 | 6 | 6
Participants | 0 | 0 | 0 | 0

11. Primary Outcome: Part 2: Number of Participants With Laboratory Values of Potential Clinical Concern
Description: Hematology parameters included hematocrit, hemoglobin, platelets, white blood cells, neutrophils, lymphocytes, monocytes, eosinophils, basophils, mean corpuscular volume, mean corpuscular hemoglobin, mean corpuscular hemoglobin concentration, red blood cells and reticulocytes. Clinical chemistry parameters included blood urea nitrogen, aspartate aminotransferase, alanine aminotransferase, gamma glutamyl transferase, alkaline phosphatase, uric acid, total protein, total and direct bilirubin, albumin, calcium, bile acids, chloride, creatinine, glucose (fasting/non-fasting), potassium, sodium and total carbon dioxide/bicarbonate. Urinalysis included specific gravity, potential of hydrogen (pH), glucose, protein, blood and ketones by dipstick and microscopic examination (within 120 minutes of collection).
Time Frame: Up to Day 22
Population: Safety Population.
Measure: Number; unit: Participants
Arm/Group | Part 2-Placebo | Part 2-Cohort B1: GSK3008356 10 mg BID (0 h, 16 h) | Part 2-Cohort B2: GSK3008356 1 mg BID (0 h, 16 h) | Part 2-Cohort B3: GSK3008356 3 mg BID (0 h, 16 h)
Number analyzed (Participants) | 6 | 6 | 6 | 6
Participants | 0 | 1 | 0 | 0

12. Primary Outcome: Part 2: Number of Participants With AE and SAE
Description: as for outcome 6
Time Frame: Up to Day 22
Population: Safety Population.
Measure: Number; unit: Participants
Arm/Group | Part 2-Placebo | Part 2-Cohort B1: GSK3008356 10 mg BID (0 h, 16 h) | Part 2-Cohort B2: GSK3008356 1 mg BID (0 h, 16 h) | Part 2-Cohort B3: GSK3008356 3 mg BID (0 h, 16 h)
Number analyzed (Participants) | 6 | 6 | 6 | 6
Participants
  AE | 3 | 5 | 6 | 5
  SAE | 0 | 0 | 0 | 0

13. Primary Outcome: Part 3: Number of Participants With Abnormal Findings in Physical Examination
Description: Part 3 was planned as a 28-day, repeat dose study in obese participants; however, since a tolerable dose with sufficient pharmacodynamic effects was not identified, this portion of the study was not conducted.
Time Frame: Up to Day 36
Population: Safety Population.
Arm/Group | Part 3: Obese Participants Cohort 1 | Part 3: Obese Participants Cohort 2 | Part 3: Obese Participants Cohort 3
Number analyzed (Participants) | 0 | 0 | 0

14. Primary Outcome: Part 3: Number of Participants With Vital Signs of Potential Clinical Concern
Description: as for outcome 13
Time Frame: Up to Day 36
Population: Safety Population.
Arm/Group | Part 3: Obese Participants Cohort 1 | Part 3: Obese Participants Cohort 2 | Part 3: Obese Participants Cohort 3
Number analyzed (Participants) | 0 | 0 | 0

15. Primary Outcome: Part 3: Number of Participants With 12-lead ECG Values of Potential Clinical Concern
Description: as for outcome 13
Time Frame: Up to Day 31
Population: Safety Population.
Arm/Group | Part 3: Obese Participants Cohort 1 | Part 3: Obese Participants Cohort 2 | Part 3: Obese Participants Cohort 3
Number analyzed (Participants) | 0 | 0 | 0

16. Primary Outcome: Part 3: Number of Participants With Clinically Significant Findings During Cardiac Monitoring
Description: as for outcome 13
Time Frame: Day 1 (Pre-dose to 4 hours post-dose)
Population: Safety Population.
Arm/Group | Part 3: Obese Participants Cohort 1 | Part 3: Obese Participants Cohort 2 | Part 3: Obese Participants Cohort 3
Number analyzed (Participants) | 0 | 0 | 0

17. Primary Outcome: Part 3: Number of Participants With Laboratory Values of Potential Clinical Concern
Description: as for outcome 13
Time Frame: Up to Day 36
Population: Safety Population.
Arm/Group | Part 3: Obese Participants Cohort 1 | Part 3: Obese Participants Cohort 2 | Part 3: Obese Participants Cohort 3
Number analyzed (Participants) | 0 | 0 | 0

18. Primary Outcome: Part 3: Number of Participants With AE and SAE
Description: as for outcome 13
Time Frame: Up to Day 36
Population: Safety Population.
Arm/Group | Part 3: Obese Participants Cohort 1 | Part 3: Obese Participants Cohort 2 | Part 3: Obese Participants Cohort 3
Number analyzed (Participants) | 0 | 0 | 0

19. Secondary Outcome: Part 1: Area Under the Concentration-time Curve (AUC) Extrapolated to Infinity (AUC[0 to Inf]), AUC From Time Zero to the Time of the Last Quantifiable Concentration (AUC[0 to t]) and AUC From Time Zero to 24 Hour (AUC[0 to 24])
Description: Blood samples for pharmacokinetic (PK) analysis of GSK3008356 were collected at the indicated time points.
Time Frame: Pre-dose, and 0.25, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 18, 24 hours post-dose on Day 1 and 36, 48, and 72 hours post-dose
Population: PK Parameter Population comprised of all participants in the PK Concentration Population (participants for whom a PK sample was obtained and analyzed) who received at least one active dose of GSK3008356 and provided PK parameters. Only those participants available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanograms/milliliters
Arm/Group | Part 1-Cohort A1: GSK3008356 5 mg | Part 1-Cohort A2: GSK3008356 10 mg | Part 1-Cohort A3: GSK3008356 30 mg | Part 1-Cohort A4: GSK3008356 75 mg | Part 1-Cohort A5: GSK3008356 200 mg | Part 1-Cohort A6: GSK3008356 125 mg | Part 1-Cohort A7: GSK3008356 100 mg (0 h, 4 h) | Part 1-Cohort A8: GSK3008356 100 mg (0 h, 16 h) | Part 1-Cohort A9: GSK3008356 200 mg Evening Dose | Part 1-Cohort A10: GSK3008356 10 mg q1h x 9 Doses | Part 1-Cohort A11: GSK3008356 5 mg q1h x 9 Doses
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 0 | 6 | 6
Hours*nanograms/milliliters
  AUC (0 to inf): number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 0 | 6 | 3
  AUC (0 to inf) | 190.004 (20.74) | 313.349 (18.23) | 840.806 (27.54) | 1960.374 (14.44) | 5493.574 (17.68) | 4042.579 (40.15) | 3364.475 (271.56) | 6018.925 (44.40) |  | 3125.413 (14.39) | 1181.752 (62.07)
  AUC (0 to t) | 184.934 (21.32) | 307.945 (17.76) | 834.100 (27.52) | 1951.059 (14.25) | 5481.127 (17.64) | 4035.511 (40.12) | 3336.805 (277.78) | 5979.430 (44.05) |  | 3121.146 (14.38) | 1246.797 (40.38)
  AUC (0 to 24): number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 0 | 6 | 3
  AUC (0 to 24) | 190.025 (20.74) | 313.369 (18.23) | 840.740 (27.54) | 1957.413 (14.11) | 5454.538 (17.24) | 4036.904 (40.09) | 3352.125 (270.66) | 5552.349 (49.03) |  | 3121.146 (14.38) | 1179.327 (61.84)

20. Secondary Outcome: Part 1: Maximum Observed Plasma Concentration (Cmax) of GSK3008356
Description: Blood samples for PK analysis of GSK3008356 were collected at the indicated time points.
Time Frame: Pre-dose, and 0.25, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 18, 24 hours post dose on Day 1 and 36, 48, and 72 hours post-dose
Population: PK Parameter Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliters
Groups:
- Part 1-Cohort A7: GSK3008356 100 mg t0, t4: Eligible participants received GSK3008356 tablets via oral route (total dose of 200 mg such that one 100 mg dose was administered at 0 h and 4 h) along with a 30% fat by calorie meal approximately 2 hours after the morning dose in a single day.
- Part 1-Cohort A8: GSK3008356 100 mg t0, t16: Eligible participants received GSK3008356 tablets via oral route (total dose of 200 mg such that one 100 mg dose was administered at 0 h and 16 h) along with a 30% fat by calorie meal approximately 2 hours after the morning dose in a single day.
Arm/Group | Part 1-Cohort A1: GSK3008356 5 mg | Part 1-Cohort A2: GSK3008356 10 mg | Part 1-Cohort A3: GSK3008356 30 mg | Part 1-Cohort A4: GSK3008356 75 mg | Part 1-Cohort A5: GSK3008356 200 mg | Part 1-Cohort A6: GSK3008356 125 mg | Part 1-Cohort A7: GSK3008356 100 mg t0, t4 | Part 1-Cohort A8: GSK3008356 100 mg t0, t16 | Part 1-Cohort A9: GSK3008356 200 mg Evening Dose | Part 1-Cohort A10: GSK3008356 10 mg q1h x 9 Doses | Part 1-Cohort A11: GSK3008356 5 mg q1h x 9 Doses
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 0 | 6 | 6
Nanograms per milliliters | 92.417 (45.40) | 190.655 (22.40) | 458.496 (33.10) | 890.913 (15.87) | 1865.337 (44.38) | 1568.035 (27.58) | 793.544 (260.32) | 946.060 (84.09) |  | 444.545 (19.61) | 202.817 (9.81)

21. Secondary Outcome: Part 1: Time to Maximum Observed Plasma Concentration (Tmax) of GSK3008356 and Apparent Terminal Half-life (t1/2) of GSK3008356
Description: Blood samples for PK analysis of GSK3008356 were collected at the indicated time points.
Time Frame: Pre-dose, and 0.25, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 18, 24 hours post dose on Day 1 and 36, 48, and 72 hours post-dose
Population: PK Parameter Population.
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Part 1-Cohort A1: GSK3008356 5 mg | Part 1-Cohort A2: GSK3008356 10 mg | Part 1-Cohort A3: GSK3008356 30 mg | Part 1-Cohort A4: GSK3008356 75 mg | Part 1-Cohort A5: GSK3008356 200 mg | Part 1-Cohort A6: GSK3008356 125 mg | Part 1-Cohort A7: GSK3008356 100 mg t0, t4 | Part 1-Cohort A8: GSK3008356 100 mg t0, t16 | Part 1-Cohort A9: GSK3008356 200 mg Evening Dose | Part 1-Cohort A10: GSK3008356 10 mg q1h x 9 Doses | Part 1-Cohort A11: GSK3008356 5 mg q1h x 9 Doses
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 0 | 6 | 6
Hours
  Tmax | 0.833 (0.4082) | 0.542 (0.2458) | 0.750 (0.2739) | 0.756 (0.2681) | 0.917 (0.5845) | 0.917 (0.5845) | 1.667 (2.1370) | 3.922 (6.9303) |  | 6.225 (3.0329) | 6.169 (2.3376)
  t1/2 | 1.501 (0.2048) | 1.425 (0.1885) | 1.623 (0.1928) | 2.113 (1.2949) | 4.545 (3.2092) | 2.779 (0.7223) | 2.540 (0.6481) | 1.752 (0.2470) |  | 1.992 (0.2050) | 1.941 (0.4058)

22. Secondary Outcome: Part 1: Cumulative Amount of Unchanged Drug Excreted Into the Urine (Ae) of GSK3008356
Description: Urine samples for PK analysis of GSK3008356 were collected at the indicated time points.
Time Frame: Pre-dose and over the post-dose intervals 0 to 12 hours and 12 to 24 hours
Population: PK Parameter Population.
Measure: Mean (Standard Deviation); unit: Nanograms*10^5
Arm/Group | Part 1-Cohort A1: GSK3008356 5 mg | Part 1-Cohort A2: GSK3008356 10 mg | Part 1-Cohort A3: GSK3008356 30 mg | Part 1-Cohort A4: GSK3008356 75 mg | Part 1-Cohort A5: GSK3008356 200 mg | Part 1-Cohort A6: GSK3008356 125 mg | Part 1-Cohort A7: GSK3008356 100 mg t0, t4 | Part 1-Cohort A8: GSK3008356 100 mg t0, t16 | Part 1-Cohort A9: GSK3008356 200 mg Evening Dose | Part 1-Cohort A10: GSK3008356 10 mg q1h x 9 Doses | Part 1-Cohort A11: GSK3008356 5 mg q1h x 9 Doses
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 0 | 6 | 6
Nanograms*10^5 | 7.958 (2.2225) | 8.699 (2.3300) | 22.738 (8.3640) | 62.332 (4.6540) | 169.051 (20.0721) | 106.273 (50.7830) | 170.777 (83.6483) | 143.269 (58.7520) |  | 91.275 (17.8857) | 28.818 (11.7506)

23. Secondary Outcome: Part 1: Renal Clearance of Drug From Plasma (CLr) of GSK3008356
Description: Urine samples for PK analysis of GSK3008356 were collected at the indicated time points.
Time Frame: Pre-dose and over the post-dose intervals 0 to 12 hours and 12 to 24 hours
Population: PK Parameter Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Milliliters per hour
Arm/Group | Part 1-Cohort A1: GSK3008356 5 mg | Part 1-Cohort A2: GSK3008356 10 mg | Part 1-Cohort A3: GSK3008356 30 mg | Part 1-Cohort A4: GSK3008356 75 mg | Part 1-Cohort A5: GSK3008356 200 mg | Part 1-Cohort A6: GSK3008356 125 mg | Part 1-Cohort A7: GSK3008356 100 mg t0, t4 | Part 1-Cohort A8: GSK3008356 100 mg t0, t16 | Part 1-Cohort A9: GSK3008356 200 mg Evening Dose | Part 1-Cohort A10: GSK3008356 10 mg q1h x 9 Doses | Part 1-Cohort A11: GSK3008356 5 mg q1h x 9 Doses
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 0 | 6 | 3
Milliliters per hour | 4115.667 (855.3612) | 2752.580 (595.2028) | 2659.878 (645.2413) | 3214.711 (539.4800) | 3091.822 (494.6096) | 2751.679 (1582.5976) | 3343.542 (765.2069) | 2638.871 (2108.5407) |  | 2935.504 (632.6009) | 1697.050 (800.8092)

24. Secondary Outcome: Part 1: Dose Proportionality of GSK3008356 for Dose 5 mg Versus (vs.) 200 mg After Single Dose Administration and Multiple Dose Administration (100 mg t0, t4 and 100 mg t0, t16) Based on AUC
Description: Dose proportionality was assessed from the AUC (0 to t) and AUC (0 to inf) obtained from multiple cohorts in Part 1. The dose proportionality was assessed using a power model on logarithmic transformation of AUC with the logarithmic transformation of dose as the single covariate in the linear regression. Point estimates and 90% confidence interval are presented.
Time Frame: Pre-dose, and 0.25, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 18, 24 hours post-dose on Day 1 and 36, 48, and 72 hours post-dose
Population: PK Parameter Population.
Measure: Number (90% Confidence Interval); unit: Slope of log dose
Groups:
- GSK3008356 5 mg, 200 mg, 100 mg 0 h, 4 h and 100 mg 0 h, 16 h: Participants received a single dose of either 5 mg or 200 mg or multiple doses of 100 mg at either 0 h and 4 h or t0 and 16 h via oral route on Day 1 of Part 1.
Arm/Group | GSK3008356 5 mg, 200 mg, 100 mg 0 h, 4 h and 100 mg 0 h, 16 h
Number analyzed (Participants) | 12
Slope of log dose
  AUC (0 to t): Cohort A5 vs. Cohort A1 | 0.92 [0.86 to 0.97]
  AUC (0 to t): Cohort A7 vs. Cohort A1 | 0.78 [0.49 to 1.08]
  AUC (0 to t): Cohort A8 vs. Cohort A1 | 0.94 [0.85 to 1.04]
  AUC (0 to inf): Cohort A5 vs. Cohort A1 | 0.91 [0.86 to 0.97]
  AUC (0 to inf): Cohort A7 vs. Cohort A1 | 0.78 [0.48 to 1.07]
  AUC (0 to inf): Cohort A8 vs. Cohort A1 | 0.94 [0.84 to 1.03]

25. Secondary Outcome: Part 1: Dose Proportionality of GSK3008356 for Dose 5 mg vs. 200 mg After Single Dose Administration Based on Cmax
Description: Dose proportionality was assessed from the Cmax obtained from multiple cohorts in Part 1. The dose proportionality was assessed using a power model on logarithmic transformation of Cmax, with the logarithmic transformation of dose as the single covariate in the linear regression. For Cmax, only a single dose group from Cohort 1 to Cohort 6 was considered since other cohorts are multiple dosing where Cmax is so different from that of single dose group. Data for Cohort A5 vs. Cohort A1 is presented, Point estimates and 90% confidence interval are presented.
Time Frame: Pre-dose, and 0.25, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 18, 24 hours post-dose on Day 1 and 36, 48, and 72 hours post-dose
Population: PK Parameter Population. Only those participants available at the specified time points were analyzed.
Measure: Number (90% Confidence Interval); unit: Slope of log dose
Groups:
- GSK3008356 5 mg and 200 mg: Participants received a single dose of either 5 mg or 200 mg via oral route on Day 1 of Part 1.
Arm/Group | GSK3008356 5 mg and 200 mg
Number analyzed (Participants) | 12
Slope of log dose | 0.81 [0.69 to 0.94]

26. Secondary Outcome: Part 1: Postprandial Triglyceride Levels Following a Single Dose and Multiple Doses of GSK3008356
Description: Preliminary pharmacodynamics of GSK3008356 was evaluated by assessing the postprandial triglyceride levels at the indicated time points. Corrected triglyceride value (Day 1) at each nominal sampling time point was defined as the corresponding post dose value by adding the following value: Part 1 Day 1 Correction: (Day -1 (1 hour + 2 hour)/2) - (Day 1 (1 hour + 2 hour)/2). Mean triglyceride levels are presented.
Time Frame: Day 1 at 1,2,3,4,5,6,7,8,9,12 hours post-dose
Population: Pharmacodynamic (PD) Population comprised of participants in the Safety population for whom at least one postprandial triglyceride sample was obtained and analyzed at Baseline and post Baseline. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Millimoles/Liters
Arm/Group | Part 1-Cohort A1: GSK3008356 5 mg | Part 1-Cohort A2: GSK3008356 10 mg | Part 1-Cohort A3: GSK3008356 30 mg | Part 1-Cohort A4: GSK3008356 75 mg | Part 1-Cohort A5: GSK3008356 200 mg | Part 1-Cohort A6: GSK3008356 125 mg | Part 1-Cohort A7: GSK3008356 100 mg t0, t4 | Part 1-Cohort A8: GSK3008356 100 mg t0, t16 | Part 1-Cohort A9: GSK3008356 200 mg Evening Dose | Part 1-Cohort A10: GSK3008356 10 mg q1h x 9 Doses | Part 1-Cohort A11: GSK3008356 5 mg q1h x 9 Doses
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 0 | 6 | 6
Millimoles/Liters
  Day 1, 1 hour post-dose | 0.925 (0.2505) | 0.900 (0.3178) | 0.800 (0.2168) | 0.767 (0.3817) | 0.742 (0.4176) | 1.008 (0.3470) | 0.717 (0.2160) | 1.242 (0.4375) |  | 0.750 (0.2588) | 0.775 (0.2842)
  Day 1, 2 hour post-dose | 0.825 (0.2505) | 0.783 (0.2733) | 0.700 (0.2168) | 0.650 (0.3317) | 0.675 (0.3283) | 0.875 (0.3029) | 0.633 (0.1992) | 1.008 (0.4913) |  | 0.667 (0.1966) | 0.692 (0.1985)
  Day 1, 3 hour post-dose | 0.825 (0.2545) | 0.817 (0.2338) | 0.717 (0.2503) | 0.667 (0.2893) | 0.592 (0.2691) | 0.842 (0.3200) | 0.750 (0.2145) | 1.042 (0.4954) |  | 0.667 (0.2066) | 0.675 (0.2162)
  Day 1, 4 hour post-dose | 1.058 (0.3056) | 0.733 (0.2273) | 0.783 (0.2805) | 0.617 (0.2696) | 0.508 (0.2538) | 0.792 (0.2333) | 0.783 (0.2910) | 0.875 (0.4084) |  | 0.600 (0.2000) | 0.592 (0.2635)
  Day 1, 5 hour post-dose | 1.308 (0.4092) | 0.867 (0.2714) | 0.950 (0.2864) | 0.767 (0.3281) | 0.558 (0.3007) | 0.825 (0.1994) | 1.000 (0.5320) | 0.958 (0.4188) |  | 0.617 (0.1780) | 0.608 (0.3024)
  Day 1, 6 hour post-dose | 1.425 (0.4612) | 0.983 (0.3531) | 1.017 (0.3502) | 0.817 (0.2582) | 0.625 (0.3126) | 0.842 (0.2836) | 1.017 (0.5663) | 1.075 (0.5223) |  | 0.700 (0.1949) | 0.642 (0.3427)
  Day 1, 7 hour post-dose | 1.275 (0.4783) | 0.967 (0.3601) | 0.950 (0.3493) | 0.850 (0.2608) | 0.658 (0.3639) | 0.842 (0.2289) | 0.917 (0.5663) | 1.175 (0.5681) |  | 0.700 (0.2098) | 0.608 (0.2923)
  Day 1, 8 hour post-dose | 1.158 (0.4018) | 0.833 (0.3093) | 0.850 (0.3464) | 0.850 (0.2000) | 0.692 (0.4104) | 0.925 (0.2444) | 0.883 (0.4782) | 1.258 (0.6078) |  | 0.670 (0.2197) | 0.592 (0.3541)
  Day 1, 9 hour post-dose | 1.008 (0.4042) | 0.750 (0.2683) | 0.733 (0.3573) | 0.767 (0.1722) | 0.675 (0.3947) | 0.858 (0.2905) | 0.850 (0.4450) | 1.292 (0.4893) |  | 0.617 (0.2714) | 0.658 (0.3484)
  Day 1, 12 hour post-dose | 0.725 (0.2697) | 0.583 (0.1693) | 0.700 (0.3178) | 0.667 (0.2090) | 0.775 (0.4263) | 0.925 (0.2525) | 0.883 (0.3173) | 1.025 (0.3984) |  | 0.700 (0.2236) | 0.792 (0.3247)

27. Secondary Outcome: Part 2: Area Under the Concentration-time Curve From Time Zero (Pre-dose) to the End of Dosing Interval (AUC[0 to Tau]) of GSK3008356 on Day 1 and Day 14
Description: Blood samples for PK analysis of GSK3008356 were collected at the indicated time points. Due to the cancellation of Part 2, Cohort B1, there are no PK parameters available on Day 14 for that dose.
Time Frame: Day 1 pre-dose, and 0.25, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 18 and 24 hours post-dose, pre-dose Day 4, 5, 6, 12 and 13 and Day 14 pre-dose, and 0.25, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 18 and 24, 36, 48 and 72 hours post dose
Population: PK Parameter Population. Only those participants available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanograms/milliliters
Arm/Group | Part 2-Cohort B1: GSK3008356 10 mg BID (0 h, 16 h) | Part 2-Cohort B2: GSK3008356 1 mg BID (0 h, 16 h) | Part 2-Cohort B3: GSK3008356 3 mg BID (0 h, 16 h)
Number analyzed (Participants) | 6 | 6 | 6
Hours*nanograms/milliliters
  AUC (0 to tau) on Day 1 | 279.222 (26.39) | 31.959 (25.16) | 107.191 (32.12)
  AUC (0 to tau) on Day 14: number analyzed (Participants) | 0 | 6 | 5
  AUC (0 to tau) on Day 14 |  | 37.429 (21.97) | 101.151 (20.20)

28. Secondary Outcome: Part 2: Cmax of GSK3008356 on Day 1 and Day 14
Description: as for outcome 27
Time Frame: as for outcome 27
Population: PK Parameter Population. Only those participants available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms/milliliters
Arm/Group | Part 2-Cohort B1: GSK3008356 10 mg BID (0 h, 16 h) | Part 2-Cohort B2: GSK3008356 1 mg BID (0 h, 16 h) | Part 2-Cohort B3: GSK3008356 3 mg BID (0 h, 16 h)
Number analyzed (Participants) | 6 | 6 | 6
Nanograms/milliliters
  Day 1 | 187.032 (28.69) | 17.638 (40.02) | 77.326 (31.73)
  Day 14: number analyzed (Participants) | 0 | 6 | 5
  Day 14 |  | 16.424 (33.86) | 46.736 (17.52)

29. Secondary Outcome: Part 2: t1/2 and Tmax of GSK3008356 on Day 1 and Day 14
Description: as for outcome 27
Time Frame: as for outcome 27
Population: PK Parameter Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Part 2-Cohort B1: GSK3008356 10 mg BID (0 h, 16 h) | Part 2-Cohort B2: GSK3008356 1 mg BID (0 h, 16 h) | Part 2-Cohort B3: GSK3008356 3 mg BID (0 h, 16 h)
Number analyzed (Participants) | 6 | 6 | 6
Hours
  t1/2 on Day 1 | 1.319 (0.1512) | 1.312 (0.1369) | 1.443 (0.1624)
  t1/2 on Day 14: number analyzed (Participants) | 0 | 6 | 5
  t1/2 on Day 14 |  | 1.406 (0.2138) | 2.115 (1.3252)
  Tmax on Day 1 | 0.517 (0.0279) | 0.583 (0.2041) | 0.436 (0.1511)
  Tmax on Day 14: number analyzed (Participants) | 0 | 6 | 5
  Tmax on Day 14 |  | 0.875 (0.6275) | 0.550 (0.2739)

30. Secondary Outcome: Part 2: Ae of GSK3008356 on Day 14
Description: Urine samples (urine concentrations or volumes) were not collected for the Part 2 of the study.
Time Frame: Pre-dose and 24 hours post-dose on Day 14
Population: PK Parameter Population.
Arm/Group | Part 2-Cohort B1: GSK3008356 10 mg BID (0 h, 16 h) | Part 2-Cohort B2: GSK3008356 1 mg BID (0 h, 16 h) | Part 2-Cohort B3: GSK3008356 3 mg BID (0 h, 16 h)
Number analyzed (Participants) | 0 | 0 | 0

31. Secondary Outcome: Part 2: CLr of GSK3008356 on Day 14
Description: Urine samples (urine concentrations or volumes) were not collected for the Part 2 of the study.
Time Frame: Pre-dose and 24 hours post-dose on Day 14
Population: PK Parameter Population.
Arm/Group | Part 2-Cohort B1: GSK3008356 10 mg BID (0 h, 16 h) | Part 2-Cohort B2: GSK3008356 1 mg BID (0 h, 16 h) | Part 2-Cohort B3: GSK3008356 3 mg BID (0 h, 16 h)
Number analyzed (Participants) | 0 | 0 | 0

32. Secondary Outcome: Part 2: Dose Proportionality of GSK3008356 for Dose 1 mg BID vs 10 mg BID and 3 mg BID After Repeat Dose Administration Based on AUC
Description: Dose proportionality was assessed from Day 1 and Day 14 AUC (0 to tau) obtained from multiple cohorts in Part 2. The dose proportionality was assessed using a power model on logarithmic transformation of AUC, with the logarithmic transformation of dose as the single covariate in the linear regression. Due to the cancellation of Part 2, Cohort B1, there are no PK parameters available on Day 14 for that dose. Point estimates and 90% confidence interval are presented.
Time Frame: as for outcome 27
Population: PK Parameter Population. Only those parameters available at the specified time points were analyzed.
Measure: Number (90% Confidence Interval); unit: Slope of log dose
Groups:
- GSK3008356 1 mg BID or 3 mg BID or 10 mg BID: Participants received multiple doses of either 1 mg BID or 3 mg BID or 10 mg BID of GSK3008356 via oral route on Day 1 and Day 14 of Part 2.
Arm/Group | GSK3008356 1 mg BID or 3 mg BID or 10 mg BID
Number analyzed (Participants) | 12
Slope of log dose
  AUC (0 to tau); Cohort B1 vs. Cohort B2 on Day 1 | 0.94 [0.83 to 1.06]
  AUC (0 to tau); Cohort B3 vs. Cohort B2 on Day 1 | 1.10 [0.83 to 1.37]
  AUC (0 to tau); Cohort B3 vs. Cohort B2 on Day 14: number analyzed (Participants) | 11
  AUC (0 to tau); Cohort B3 vs. Cohort B2 on Day 14 | 0.90 [0.69 to 1.12]
  AUC (0 to inf); Cohort B1 vs. Cohort B2 on Day 1 | 0.94 [0.83 to 1.06]
  AUC (0 to inf); Cohort B3 vs. Cohort B2 on Day 1 | 1.10 [0.83 to 1.37]

33. Secondary Outcome: Part 2: Dose Proportionality of GSK3008356 for Dose 1 mg BID vs 10 mg BID and 3 mg BID After Repeat Dose Administration Based on Cmax
Description: The dose proportionality was assessed using a power model on logarithmic transformation of Cmax, with the logarithmic transformation of dose as the single covariate in the linear regression. Due to the cancellation of Part 2, Cohort B1, there are no PK parameters available on Day 14 for that dose. Point estimates and 90% confidence interval are presented for Day 1 and Day 14 of Part 2.
Time Frame: Day 1 pre-dose, and 0.25, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 18 and 24 hours post-dose, pre-dose Day 4, 5, 6, 12 and 13 and Day 14 pre-dose, and 0.25, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 18 and 24, 36, 48 and 72 hours post-dose
Population: PK Parameter Population.
Measure: Number (90% Confidence Interval); unit: Slope of log dose
Arm/Group | GSK3008356 1 mg BID or 3 mg BID or 10 mg BID
Number analyzed (Participants) | 12
Slope of log dose
  Cmax; Cohort B1 vs. Cohort B2 on Day 1 | 1.03 [0.87 to 1.18]
  Cmax; Cohort B3 vs. Cohort B2 on Day 1 | 1.35 [1.01 to 1.68]
  Cmax; Cohort B3 vs. Cohort B2 on Day 14: number analyzed (Participants) | 11
  Cmax; Cohort B3 vs. Cohort B2 on Day 14 | 0.95 [0.68 to 1.23]

34. Secondary Outcome: Part 2: Observed Accumulation Ratio of GSK3008356
Description: Observed accumulation ratio based on AUC(0- tau) is (Ro), and based on Cmax is (RCmax). Ro was calculated as the ratio [AUC0-tau on the final day (Day 14)]/[ AUC0-tau on Day 1] and Rcmax was calculated as the ratio [Cmax on the final day (Day 14)]/[Cmax on Day 1]. Blood samples for PK analysis of GSK3008356 were collected at the indicated time points.
Time Frame: as for outcome 27
Population: PK Parameter Population. Only those participants available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Part 2-Cohort B1: GSK3008356 10 mg BID (0 h, 16 h) | Part 2-Cohort B2: GSK3008356 1 mg BID (0 h, 16 h) | Part 2-Cohort B3: GSK3008356 3 mg BID (0 h, 16 h)
Number analyzed (Participants) | 0 | 6 | 5
Ratio
  Ro |  | 1.171 (13.52) | 1.010 (19.76)
  Rcmax |  | 0.931 (22.64) | 0.606 (38.82)

35. Secondary Outcome: Part 2: Trough Plasma Concentrations (Ctrough) to Assess Steady State of GSK3008356 Following 14-day Repeat Dosing
Description: Ctrough is the observed concentration at the end of a dosing interval, immediately before next administration. Due to the cancellation of Part 2, Cohort B1, there are no PK parameters available on Day 14 for that dose.
Time Frame: Pre-dose on Days 2, 4, 5, 6, 12, 13, 14 and the 24 hours post-dose on Day 14
Population: PK Parameter Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Nanograms/Milliliters
Arm/Group | Part 2-Cohort B1: GSK3008356 10 mg BID (0 h, 16 h) | Part 2-Cohort B2: GSK3008356 1 mg BID (0 h, 16 h) | Part 2-Cohort B3: GSK3008356 3 mg BID (0 h, 16 h)
Number analyzed (Participants) | 6 | 6 | 6
Nanograms/Milliliters
  Day 1, 24 Hour | 11.953 (7.8239) | 2.595 (2.0718) | 4.025 (1.7353)
  Day 4, Pre-Dose: number analyzed (Participants) | 4 | 6 | 6
  Day 4, Pre-Dose | 11.528 (7.2515) | 1.362 (0.7706) | 1.940 (2.2364)
  Day 5, Pre-Dose: number analyzed (Participants) | 4 | 6 | 6
  Day 5, Pre-Dose | 4.790 (2.2425) | 1.392 (1.6697) | 6.595 (4.8009)
  Day 6, Pre-Dose: number analyzed (Participants) | 3 | 6 | 6
  Day 6, Pre-Dose | 2.880 (2.6985) | 0.475 (0.7364) | 3.206 (1.9157)
  Day 12, Pre-Dose: number analyzed (Participants) | 0 | 6 | 5
  Day 12, Pre-Dose |  | 0.205 (0.5021) | 1.934 (1.0154)
  Day 13, Pre-Dose: number analyzed (Participants) | 0 | 6 | 5
  Day 13, Pre-Dose |  | 0.325 (0.7961) | 3.756 (2.1434)
  Day 14, Pre-Dose: number analyzed (Participants) | 0 | 6 | 5
  Day 14, Pre-Dose |  | 1.587 (1.3835) | 4.368 (3.3806)
  Day 14, 24 Hour: number analyzed (Participants) | 0 | 6 | 5
  Day 14, 24 Hour |  | 1.420 (0.6255) | 1.866 (0.4191)

36. Secondary Outcome: Part 2: Postprandial Triglyceride Levels Following 14-day Repeat Dosing of GSK3008356
Description: Preliminary pharmacodynamics of GSK3008356 was evaluated by assessing the postprandial triglyceride levels at the indicated time points. Corrected TG value (Day 1 and Day 14) at each nominal sampling time point defined as the corresponding post dose value by adding the following value: Part 2 Day 1 Correction: (Day -1 (1 hour + 2 hour)/2) - (Day 1 (1 hour + 2 hour)/2); Part 2 Day 14 Correction: (Day -1 (1 hour + 2 hour)/2) - (Day 14 (1 hour + 2 hour)/2). Mean triglyceride levels are presented.
Time Frame: Day 1 (1, 2, 3, 4, 5, 6, 7, 8, 9 and 12 hours post-dose) and Day 14 (1, 2, 3, 4, 5, 6, 7, 8, 9 and 12 hours post-dose)
Population: PD Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Millimoles/Liter
Arm/Group | Part 2-Cohort B1: GSK3008356 10 mg BID (0 h, 16 h) | Part 2-Cohort B2: GSK3008356 1 mg BID (0 h, 16 h) | Part 2-Cohort B3: GSK3008356 3 mg BID (0 h, 16 h)
Number analyzed (Participants) | 6 | 6 | 6
Millimoles/Liter
  Day 1, 1 hour post-dose | 0.867 (0.4987) | 0.950 (0.3017) | 1.217 (0.3697)
  Day 1, 2 hour post-dose | 0.800 (0.4219) | 0.783 (0.2317) | 0.950 (0.2236)
  Day 1, 3 hour post-dose | 0.767 (0.4987) | 0.883 (0.3189) | 0.983 (0.2503)
  Day 1, 4 hour post-dose | 0.883 (0.4956) | 0.833 (0.3235) | 1.067 (0.3220)
  Day 1, 5 hour post-dose | 1.033 (0.4633) | 1.017 (0.4309) | 1.317 (0.4655)
  Day 1, 6 hour post-dose | 1.150 (0.4990) | 1.050 (0.6189) | 1.500 (0.5523)
  Day 1, 7 hour post-dose | 1.300 (0.5933) | 1.233 (0.7005) | 1.700 (0.3987)
  Day 1, 8 hour post-dose | 1.283 (0.7561) | 1.167 (0.6578) | 1.717 (0.4676)
  Day 1, 9 hour post-dose | 1.050 (0.6442) | 1.000 (0.6293) | 1.467 (0.5037)
  Day 1, 12 hour post-dose | 0.800 (0.4359) | 0.717 (0.3996) | 1.033 (0.2041)
  Day 14, 1 hour post-dose: number analyzed (Participants) | 0 | 6 | 5
  Day 14, 1 hour post-dose |  | 0.917 (0.3077) | 1.020 (0.2490)
  Day 14, 2 hour post-dose: number analyzed (Participants) | 0 | 6 | 5
  Day 14, 2 hour post-dose |  | 0.817 (0.2582) | 0.960 (0.1597)
  Day 14, 3 hour post-dose: number analyzed (Participants) | 0 | 6 | 5
  Day 14, 3 hour post-dose |  | 0.950 (0.2757) | 1.080 (0.1924)
  Day 14, 4 hour post-dose: number analyzed (Participants) | 0 | 6 | 5
  Day 14, 4 hour post-dose |  | 1.017 (0.2840) | 1.020 (0.2907)
  Day 14, 5 hour post-dose: number analyzed (Participants) | 0 | 6 | 5
  Day 14, 5 hour post-dose |  | 1.100 (0.3860) | 1.060 (0.2748)
  Day 14, 6 hour post-dose: number analyzed (Participants) | 0 | 6 | 5
  Day 14, 6 hour post-dose |  | 1.217 (0.5066) | 1.260 (0.3943)
  Day 14, 7 hour post-dose: number analyzed (Participants) | 0 | 6 | 5
  Day 14, 7 hour post-dose |  | 1.367 (0.5345) | 1.460 (0.2608)
  Day 14, 8 hour post-dose: number analyzed (Participants) | 0 | 6 | 5
  Day 14, 8 hour post-dose |  | 1.367 (0.4834) | 1.380 (0.4764)
  Day 14, 9 hour post-dose: number analyzed (Participants) | 0 | 6 | 5
  Day 14, 9 hour post-dose |  | 0.817 (0.4844) | 1.220 (0.5239)
  Day 14, 12 hour post-dose: number analyzed (Participants) | 0 | 6 | 5
  Day 14, 12 hour post-dose |  | 0.800 (0.4889) | 0.720 (0.6079)

37. Secondary Outcome: Part 3: AUC (0-tau) of GSK3008356 on Day 1 and Day 28
Description: as for outcome 13
Time Frame: Pre-dose, 0.25, 0.5, 1, 1.5, 2, 4, 6, 8 (only in cohort 1), 12, 14 (only in cohorts 2 and 3), 18, and 24 hours post-dose on Day 1 and Day 28 and additionally 36, 48, and 72 hours post-dose on Day 28
Population: PK Parameter Population.
Arm/Group | Part 3: Obese Participants Cohort 1 | Part 3: Obese Participants Cohort 2 | Part 3: Obese Participants Cohort 3
Number analyzed (Participants) | 0 | 0 | 0

38. Secondary Outcome: Part 3: Cmax of GSK3008356 on Day 1 and Day 28
Description: as for outcome 13
Time Frame: as for outcome 37
Population: PK Parameter Population.
Arm/Group | Part 3: Obese Participants Cohort 1 | Part 3: Obese Participants Cohort 2 | Part 3: Obese Participants Cohort 3
Number analyzed (Participants) | 0 | 0 | 0

39. Secondary Outcome: Part 3: Tmax of GSK3008356 on Day 1 and Day 28
Description: as for outcome 13
Time Frame: as for outcome 37
Population: PK Parameter Population.
Arm/Group | Part 3: Obese Participants Cohort 1 | Part 3: Obese Participants Cohort 2 | Part 3: Obese Participants Cohort 3
Number analyzed (Participants) | 0 | 0 | 0

40. Secondary Outcome: Part 3: t1/2 of GSK3008356 on Day 28
Description: as for outcome 13
Time Frame: Pre-dose, 0.25, 0.5, 1, 1.5, 2, 4, 6, 8 (only in cohort 1), 12, 14 (only in cohorts 2 and 3), 18, 24, 36, 48, and 72 hours post-dose on Day 28
Population: PK Parameter Population.
Arm/Group | Part 3: Obese Participants Cohort 1 | Part 3: Obese Participants Cohort 2 | Part 3: Obese Participants Cohort 3
Number analyzed (Participants) | 0 | 0 | 0

41. Secondary Outcome: Part 3: Ae of GSK3008356 on Day 28
Description: as for outcome 13
Time Frame: Day 28 in each cohort
Population: PK Parameter Population.
Arm/Group | Part 3: Obese Participants Cohort 1 | Part 3: Obese Participants Cohort 2 | Part 3: Obese Participants Cohort 3
Number analyzed (Participants) | 0 | 0 | 0

42. Secondary Outcome: Part 3: CLr of GSK3008356 on Day 28
Description: as for outcome 13
Time Frame: Day 28 in each cohort
Population: PK Parameter Population.
Arm/Group | Part 3: Obese Participants Cohort 1 | Part 3: Obese Participants Cohort 2 | Part 3: Obese Participants Cohort 3
Number analyzed (Participants) | 0 | 0 | 0

43. Secondary Outcome: Part 3: Dose Proportionality of GSK3008356
Description: as for outcome 13
Time Frame: Pre-dose, 0.25, 0.5, 1, 1.5, 2, 4, 6, 8 (only in cohort 1), 12, 14 (only in cohorts 2 and 3), 18, and 24 hours post-dose on Days 1 and 28 and additionally 36, 48, and 72 hours post-dose on Day 28
Population: PK Parameter Population.
Groups:
- Part 3: Cohort 1 to Cohort 3: Participants in this arm were planned to receive 28 daily doses so as to evaluate 1 dose strength of GSK3008356 administered as morning doses.
Arm/Group | Part 3: Cohort 1 to Cohort 3
Number analyzed (Participants) | 0

44. Secondary Outcome: Part 3: Observed Accumulation Ratio of GSK3008356
Description: as for outcome 13
Time Frame: as for outcome 43
Population: PK Parameter Population.
Arm/Group | Part 3: Obese Participants Cohort 1 | Part 3: Obese Participants Cohort 2 | Part 3: Obese Participants Cohort 3
Number analyzed (Participants) | 0 | 0 | 0

45. Secondary Outcome: Part 3: Ctrough to Assess Steady State of GSK3008356 Following 28-day Repeat Dosing
Description: as for outcome 13
Time Frame: as for outcome 43
Population: PK Parameter Population.
Arm/Group | Part 3: Obese Participants Cohort 1 | Part 3: Obese Participants Cohort 2 | Part 3: Obese Participants Cohort 3
Number analyzed (Participants) | 0 | 0 | 0

46. Secondary Outcome: Part 3: Postprandial Triglyceride Levels Following 28-day Repeat Dosing of GSK3008356 in Obese Participants
Description: as for outcome 13
Time Frame: Day -1, Day 1, and Day 28 in cohort 1, and Day 1, Day 2, and Day 28 in cohorts 2 and 3
Population: PD Population.
Arm/Group | Part 3: Obese Participants Cohort 1 | Part 3: Obese Participants Cohort 2 | Part 3: Obese Participants Cohort 3
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Serious adverse events and non-serious adverse events were collected from the start of study treatment until the follow-up contact (Up to 8 days for Part 1 and up to 22 days for Part 2)
Description: Serious adverse events and non-serious adverse events were collected for the Safety Population which comprised of all participants who received at least one dose of study medication. Non-serious adverse events and serious adverse events were not collected in Part 3 as no participants were enrolled. All non-serious adverse events with a frequency threshold of more than 3 occurrences in any part is presented.
Arm/Group | Part 1- Placebo | Part 1-Cohort A1: GSK3008356 5 mg | Part 1-Cohort A2: GSK3008356 10 mg | Part 1-Cohort A3: GSK3008356 30 mg | Part 1-Cohort A4: GSK3008356 75 mg | Part 1-Cohort A5: GSK3008356 200 mg | Part 1-Cohort A6: GSK3008356 125 mg | Part 1-Cohort A7: GSK3008356 100 mg BID (0 h, 4 h) | Part 1-Cohort A8: GSK3008356 100 mg BID (0 h, 16 h) | Part 1-Cohort A9: GSK3008356 200 mg Evening Dose | Part 1-Cohort A10: GSK3008356 10 mg q1h x 9 Doses | Part 1-Cohort A11: GSK3008356 5 mg q1h x 9 Doses | Part 2-Placebo | Part 2-Cohort B1: GSK3008356 10 mg BID (0 h, 16 h) | Part 2-Cohort B2: GSK3008356 1 mg BID (0 h, 16 h) | Part 2-Cohort B3: GSK3008356 3 mg BID (0 h, 16 h) | Part 3: Obese Participants Cohort 1 | Part 3: Obese Participants Cohort 2 | Part 3: Obese Participants Cohort 3
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/0 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/0 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/20 | 1/6 | 0/6 | 1/6 | 1/6 | 3/6 | 3/6 | 3/6 | 3/6 | 0/0 | 0/6 | 3/6 | 2/6 | 5/6 | 3/6 | 3/6 | 0/0 | 0/0 | 0/0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1- Placebo (N=20) | Part 1-Cohort A1: GSK3008356 5 mg (N=6) | Part 1-Cohort A2: GSK3008356 10 mg (N=6) | Part 1-Cohort A3: GSK3008356 30 mg (N=6) | Part 1-Cohort A4: GSK3008356 75 mg (N=6) | Part 1-Cohort A5: GSK3008356 200 mg (N=6) | Part 1-Cohort A6: GSK3008356 125 mg (N=6) | Part 1-Cohort A7: GSK3008356 100 mg BID (0 h, 4 h) (N=6) | Part 1-Cohort A8: GSK3008356 100 mg BID (0 h, 16 h) (N=6) | Part 1-Cohort A9: GSK3008356 200 mg Evening Dose (N=0) | Part 1-Cohort A10: GSK3008356 10 mg q1h x 9 Doses (N=6) | Part 1-Cohort A11: GSK3008356 5 mg q1h x 9 Doses (N=6) | Part 2-Placebo (N=6) | Part 2-Cohort B1: GSK3008356 10 mg BID (0 h, 16 h) (N=6) | Part 2-Cohort B2: GSK3008356 1 mg BID (0 h, 16 h) (N=6) | Part 2-Cohort B3: GSK3008356 3 mg BID (0 h, 16 h) (N=6) | Part 3: Obese Participants Cohort 1 (N=0) | Part 3: Obese Participants Cohort 2 (N=0) | Part 3: Obese Participants Cohort 3 (N=0)
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 5 | 3 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 2 | 2 | 4 | 1 | 3 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 1 | 2 | 0 | 0 | 1 | 1 | 3 | 1 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2017-02-07): https://cdn.clinicaltrials.gov/large-docs/66/NCT02742766/Prot_000.pdf
  • Statistical Analysis Plan (2017-08-03): https://cdn.clinicaltrials.gov/large-docs/66/NCT02742766/SAP_001.pdf